CLINICAL TRIAL: NCT03692676
Title: Characteristics of Patients Initiating Spiriva Respimat in Asthma in the UK: a Cross-sectional Study Based on the Clinical Practice Research Datalink
Brief Title: Characteristics of Pts Initiating Spiriva Respimat in Asthma
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0205-0537
Record Dates: First submitted 2018-09-25; First posted 2018-10-02 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects with Asthma: Asthmatic patients prescribed Inhaled corticosteroids/Long-acting beta agonists (ICS/LABA FDC) before index date, initiated with Spiriva Respimat, or received a higher dose of ICS/LABA FDC, initiated LTRA , or switched to a new ICS/LABA FDC fom the previous ICS/LABA FDC
  Interventions: Device: Spiriva Respimat

INTERVENTIONS:
Device: Spiriva Respimat — soft-mist inhaler

SUMMARY:
This study is a cross-sectional, non-interventional study based on existing data (NISed).

DETAILED DESCRIPTION:
The UK CPRD data will be used to assess the characteristics of asthma patients who were prescribed ICS/LABA FDC before the index date and who initiated Spiriva Respimat, or received a higher dose of ICS/LABA FDC, or initiated LTRA, or switched to a new ICS/LABA FDC in the UK during the study period (September 2014-December 2017) enabling to assess potential channeling of prescribing to different patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above at the index date
* At least 12 months of continuous registration prior to the index date in a practice contributing up to standard (UTS) data to the Clinical Practice Research Database (CPRD)
* Had a diagnosis of asthma before the index date
* Being treated with Inhaled corticosteroids/Long-acting beta agonists (ICS LABA FDC) before the index date (at least one prescription within 3 months before the index date)
* Patients who were new users of Spiriva Respimat, or LTRA, or patients who were prescribed a higher dose of ICS/LABA FDC, or patients who switched to a new ICS/LABA FDC from the previous ICS/LABA FDC

Exclusion Criteria:

* Patients who were prescribed other Long-acting muscarinic antagonists (LAMA) any time before or on the index date
* In the primary analysis, patients who were diagnosed with COPD before or on the index date will be excluded from the study. In a sensitivity analysis, patients who had both asthma and COPD diagnoses will be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic patients who were prescribed ICS/LABA FDC before the index date and who initiated Spiriva Respimat, or received a higher dose of ICS/LABA FDC, or initiated LTRA, or switched to a new ICS/LABA FDC from the previous ICS/LABA FDC in the UK during the study period (September, 2014-December 31, 2017)
Sampling Method: Non-Probability Sample
Enrollment: 116133 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim, Ingelheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is a cross-sectional assessment of asthma patients who initiated Spiriva Respimat, who initiated leukotriene receptor antagonist (LTRA), who received a higher dose of ICS/LABA FDC, or who switched to a new ICS/LABA FDC in asthma in the UK during the study period (September, 2014-December 31, 2017). (Non-interventional study based on existing data).
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects meeting the exclusion criteria were excluded.
Groups:
- Spiriva Respimat: The first Spiriva Respimat prescription record during study period qualifies for cohort entry and its event date will be set as index date.
  Patients will be excluded if they fulfill any of the following exclusion criteria:
  * prior Spiriva Respimat use before index date
  * no Inhaled corticosteroids (ICS)/ Long-acting beta agonists (LABA) Fixed Dose Combination (FDC) Prescription Record (Rx) within 3 months before index date
  * no prior asthma Diagnosis Record (Dx) before index date
  * age on index date less than 18 years
  * on index date less than 365 days prior Up-to-standard (UTS) registration
  * prior Chronic Obstructive Pulmonary Disease (COPD) Dx before index date (including index date)
  * any prior Long-acting muscarinic antagonists (LAMA) use (including index date)
- Leukotriene Receptor Antagonist (LTRA): The first LTRA prescription record during study period qualifies for cohort entry and its event date will be set as index date.
  Patients will be excluded if they fulfill any of the following exclusion criteria:
  * prior LTRA use before index date
  * no ICS/LABA FDC Rx within 3 months before index date
  * no prior asthma Dx before index date age on index date less than 18 years
  * on index date less than 365 days prior UTS registration
  * prior COPD Dx before index date (including index date)
  * any prior LAMA use before index date (including index date)
- ICS/LABA Fixed Dose Combination (Switchers): The first ICS/LABA FDC prescription record during study period with different ICS and/or LABA drug substance component as compared to the preceding FDC prescription qualifies for cohort entry and its event date will be set as index date. Same ICS/LABA FDC, but different device (e.g. switch from DPI to pMDI) will trigger cohort entry to this cohort as well.
  Patients will be excluded if they fulfil any of the following exclusion criteria:
  * prior use of the same ICS/LABA FDC (evaluated on drug substance and device level) before index date
  * preceding ICS/LABA FDC Rx not within 3 months before index date
  * no prior asthma Dx before index date
  * age on index date less than 18 years
  * on index date less than 365 days prior UTS registration
  * prior COPD Dx before index date (including index date)
  * any prior LAMA use before index date (including index date)
- ICS Dose Increase of ICS/LABA Fixed Dose Combination User: The first ICS/LABA FDC prescription record during study period which represent a dose increase of ICS daily dose as compared to the preceding FDC prescription qualifies for cohort entry and its event date will be set as index date.
  Patients will be excluded if they fulfill any of the following exclusion criteria:
  * preceding ICS/LABA FDC Rx within 3 months before index date
  * no prior asthma Dx before index date
  * age on index date less than 18 years
  * on index date less than 365 days prior UTS registration
  * prior COPD Dx before index date (incl. index date)
  * any prior LAMA use before index date (incl. index date)
Period: Overall Study
Arm/Group | Spiriva Respimat | Leukotriene Receptor Antagonist (LTRA) | ICS/LABA Fixed Dose Combination (Switchers) | ICS Dose Increase of ICS/LABA Fixed Dose Combination User
Started | 10365 | 51142 | 49479 | 5147
Completed | 940 | 3704 | 11135 | 1561
Not Completed | 9425 | 47438 | 38344 | 3586
Not completed — exclude patients with prior use | 4424 | 24726 | 0 | 0
Not completed — exclude patients without concurrent ICS/LABA FDC use | 2480 | 19037 | 0 | 0
Not completed — exclude patients without prior recorded asthma diagnosis | 881 | 563 | 6281 | 558
Not completed — exclude patients less than 18 years of age on index date | 8 | 613 | 836 | 193
Not completed — exclude patients with less than 1 year prior continous UTS enrollment | 149 | 717 | 1723 | 273
Not completed — exclude patients with prior LAMA use (any time prior to index date) | 1208 | 759 | 7419 | 684
Not completed — exclude patients with prior recorded COPD diagnosis | 275 | 218 | 1515 | 173
Not completed — exclude patients with multiple FDC prescriptions on index date | 0 | 0 | 1147 | 4
Not completed — exclude patients with prior use of same substances and device | 0 | 0 | 3700 | 0
Not completed — exclude patients without ICS/LABA FDC prescription within 3 months prior to index date | 0 | 0 | 14965 | 1198
Not completed — exclude patients with different substance(s)/device at preceding prescription | 0 | 0 | 0 | 223
Not completed — Other | 0 | 805 | 758 | 277
Not completed — exclude patients with multiple substance(s)/device at preceding prescription | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Asthma patients who initiated Spiriva Respimat, who initiated leukotriene receptor antagonist (LTRA), who received a higher dose of ICS/LABA FDC, or who switched to a new ICS/LABA FDC in asthma, and who did not violate any of the exclusion criteria, in the United Kingdom during the study period (Sep 2014 - Dec 2017).
Groups:
- Total: Total of all reporting groups
Arm/Group | Spiriva Respimat | Leukotriene Receptor Antagonist (LTRA) | ICS/LABA Fixed Dose Combination (Switchers) | ICS Dose Increase of ICS/LABA Fixed Dose Combination User | Total
Number analyzed (Participants) | 940 | 3704 | 11135 | 1561 | 17340
Age, Continuous [Mean (Standard Deviation); unit: Year] | 54.22 (15.741) | 49.12 (16.299) | 53.31 (16.961) | 51.91 (17.189) | 52.34 (16.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 653 | 2479 | 7121 | 979 | 11232
  Male | 287 | 1225 | 4014 | 582 | 6108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 25 | 90 | 210 | 42 | 367
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 30 | 71 | 9 | 119
  White | 527 | 1996 | 5896 | 776 | 9195
  More than one race | 13 | 40 | 99 | 14 | 166
  Unknown or Not Reported | 366 | 1548 | 4859 | 720 | 7493

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cardiac Arrhythmias
Description: The number of participants who had Cardiac arrhythmias on the index date or in the year prior to the index date.
Time Frame: On the index date or in the year prior to the index date
Population: Asthma patients who initiated Spiriva Respimat, who initiated leukotriene receptor antagonist (LTRA), who received a higher dose of ICS/LABA FDC, or who switched to a new ICS/LABA FDC in asthma, and who did not violate any of the exclusion criteria, in the United Kingdom during the studied period (Sep 2014 - Dec 2017).
Measure: Count of Participants; unit: Participants
Arm/Group | Spiriva Respimat | Leukotriene Receptor Antagonist (LTRA) | ICS/LABA Fixed Dose Combination (Switchers) | ICS Dose Increase of ICS/LABA Fixed Dose Combination User
Number analyzed (Participants) | 940 | 3704 | 11135 | 1561
Participants | 11 | 17 | 102 | 16

2. Secondary Outcome: Number of Participants With Cardiac Failure
Description: The number of participants who had Cardiac failure on the index date or in the year prior to the index date.
Time Frame: On the index date or in the year prior to the index date
Population: as for outcome 1
Measure: Number; unit: Patients with cardiac failures
Arm/Group | Spiriva Respimat | Leukotriene Receptor Antagonist (LTRA) | ICS/LABA Fixed Dose Combination (Switchers) | ICS Dose Increase of ICS/LABA Fixed Dose Combination User
Number analyzed (Participants) | 940 | 3704 | 11135 | 1561
Patients with cardiac failures | NA — NA = <5, for compliance with Independent Scientific Advisory Committee (ISAC) requirements, any covariate resulting in counts less than 5 will be reported as "<5" without any further reporting. | 9 | 49 | 12

ADVERSE EVENTS:
Time Frame: In this non-interventional study based on existing data, All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: In this non-interventional study based on existing data, All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Spiriva Respimat | Leukotriene Receptor Antagonist (LTRA) | ICS/LABA Fixed Dose Combination (Switchers) | ICS Dose Increase of ICS/LABA Fixed Dose Combination User
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT03692676/Prot_002.pdf
  • Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03692676/SAP_003.pdf